CLINICAL TRIAL: NCT05604677
Title: Factors Influencing the Decision-making Process for Breast Surgery in Women Likely to Face Breast Cancer.
Brief Title: Factor Influencing Breast Surgery Type Decision-Making
Status: Completed | Type: Observational
Sponsor: Etienne El Helou (Other)
Responsible Party: Sponsor-Investigator, Etienne El Helou, Principal Investigator, Dr Etienne El Helou
Organization: Dr Etienne El Helou (Other)
Other Study IDs: HelouEl
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Mastectomy; Breast Conserving Surgery; Lebanese Population; Surgical Choice; Oncoplastic Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast Surgery — Breast-conserving Surgery or modified radical mastectomy

SUMMARY:
The aim of this observational study is to determine the factors influencing the decision-making process for breast surgery type, in Lebanese women likely to face breast cancer.

The main questions it aims to answer are the presence or not of a correlation between the type of choice and the following data:

* Demographic
* Health Status
* Several factors that may influence the decision

Participants will complete a well-structured and organized online survey

ELIGIBILITY:
Inclusion Criteria:

* Lebanese Females

Exclusion Criteria:

* None

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Lebanese Females
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Influencing Factors | 2 months
  Factors influencing breast surgery type decision making process

CONTACTS AND LOCATIONS:
Overall Officials: Etienne El-Helou, MD, Principal Investigator — Dr Etienne El Helou
Locations (1):
- HelouEl, Baabda, Mount Lebanon, Lebanon